CLINICAL TRIAL: NCT01065818
Title: Early Prediction of Pathology Response of Chemoradiotherapy With FLT PET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAD5444; R21CA121551 (NIH)
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-08

CONDITIONS: Esophageal Cancer; Non-small Cell Lung Cancer
Keywords: Esophageal cancer; Non-small cell lung cancer; FLT-PET; Chemoradiotherapy
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fluoro-L-Thymidine (Experimental): Injection pre-Neoadjuvant Therapy (CRT, CT, or RT) and post-3 weeks Neoadjuvant Therapy (CRT, CT, RT)(3 weeks from the start of Neoadjuvant Therapy) prior to surgery.
  Interventions: Drug: Fluoro-L-Thymidine

INTERVENTIONS:
Drug: Fluoro-L-Thymidine — 4D-PET/CT imaging with an injection of Fluoro-L-Thymidine at pre-Neoadjuvant Therapy and post-3 weeks Neoadjuvant Therapy prior to surgery.
  Other Names: FLT

SUMMARY:
The goal of this research study is to learn if a new type of PET scan (18F-FLT) can help to better detect changes of tumor growth rate (or how active) in esophagus cancer and lung cancer Researchers will study at what time during treatment the 18F-FLT PET scan should be given to get the best results. A Positron Emission Tomography (PET) scan is a type of scan that uses a radioactive solution to locate cancer cells inside the body. Using the PET scan, doctors can locate solid tumors and collect information about how "active" the cancer cells are. For this study, a new type of solution, [F-18]-ﬂuoro-L-thymidine (FLT), will be used. FLT can detect actively growing tumor, and researchers hope that FLT may be able to help provide information about how well esophagus cancer treatment is working. This information could be used to help predict if the cancer will respond to treatment.

All enrolled subjects will receive PET/CT imaging at pre-Neoadjuvant Therapy and post-3 weeks Neoadjuvant Therapy (3 weeks from the start of Neoadjuvant Therapy) prior to the surgery. At each time of the PET/CT procedure, the subject will receive an injection of FLT which is an investigational pharmaceutical labeled with radioactive ﬂuorine. 45-60 mines after the FLT injection, the scan will be performed. Each scan might take 10-15 minutes. Participation in this pilot study will not change the patients normal chemotherapy, radiation treatment, and surgery recommended the patients physician as parts of their standard of care.

DETAILED DESCRIPTION:
The goal of the study is to obtain preliminary data and initial estimates of the FLT ability-PET to identify pathCR patients who have esophageal carinoma or non-small cell lung cancer and undergo Neoadjuvant Therapy (Chemoradiotherapy, Chemotherapy or Radiation Therapy) prior to surgery. Achievement in pathCR after pre-operative Neoadjuvant Therapy is associated with improved patient outcomes; however, there is no effective method to predict pathological response before surgery. Thus, a patient with pathCR , for whom esophagectomy or thoracoscopy may be unnecessary, still undergoes surgery and faces the prohibitive side effects of this surgical procedure. Additionally, Neoadjuvant Therapy is associated with considerable morbidities and tool to predict and avoid ineffective therapy are lacking. Because deregulated proliferation is one of the hallmarks of cancer and its proliferation rate is associated with aggressive biologic behavior and response to therapy, imaging the proliferative state of cancer cells by non-invasive functional imaging is of great interest. Recently 18F-FLT (3'deoxy33'-18F- ﬂuorothymidine) has been reported as a promising PET radiopharmaceutical for imaging cancer proliferation and has been validated in several in vitro & in vivo models. However, only a few studies addressed its role in depicting changes in cancer proliferation and assessing response to Neoadjuvant Therapy, and none of these studies have focused on esophageal cancer and lung cancer. We propose to conduct a pilot study to learn the optimal FLT PET imaging timepoint during the early course of Neoadjuvant Therapy that has the highest predictive value for pathCR in patients with esophageal cancer or lung cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients with histologically diagnosed adenocarcinoma or squamous cell carcinoma of the esophagus and locoregional disease (stages II and III) and locally advanced non-small cell lung cancer (stage III) will be eligible for participation in this study.

Exclusion Criteria:

* Abnormal liver function (<2.5 x ULN of aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ; <1.5 x upper limit of normal (ULN) of bilirubin total) or abnormal renal function (<1.5 x ULN of creatinine) or peripheral neuropathy
* Women with pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K.S. Clifford Chao, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluoro-L-Thymidine: Injection pre-Neoadjuvant Therapy (CRT, CT, or RT) and post-3 weeks Neoadjuvant Therapy (CRT, CT, RT)(3 weeks from the start of Neoadjuvant Therapy) prior to surgery.
  Fluoro-L-Thymidine (FLT): 4-dimensional (4D)-Positron Emission Tomography (PET)/CT imaging with an injection of Fluoro-L-Thymidine at pre-Neoadjuvant Therapy and post-3 weeks Neoadjuvant Therapy prior to surgery.
Period: Overall Study
Arm/Group | Fluoro-L-Thymidine
Started | 6
Completed | 4
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Not a candidate for surgery | 1

BASELINE CHARACTERISTICS:
Groups:
- Fluoro-L-Thymidine: Injection pre-Neoadjuvant Therapy (CRT, CT, or RT) and post-3 weeks Neoadjuvant Therapy (CRT, CT, RT)(3 weeks from the start of Neoadjuvant Therapy) prior to surgery.
  Fluoro-L-Thymidine: 4D-PET/CT imaging with an injection of Fluoro-L-Thymidine at pre-Neoadjuvant Therapy and post-3 weeks Neoadjuvant Therapy prior to surgery.
  Data on age (per age categories) and race/ethnicity was not available for these 6 subjects. Only sex was available.
Arm/Group | Fluoro-L-Thymidine
Number analyzed (Participants) | 6
Age, Customized [Count of Participants; unit: Participants]
  >18 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Optimal Timepoint During the Course of Neoadjuvant Therapy [CRT, CT (Chemotherapy) or RT Radiotherapy)] That FLT-PET Imaging Can Predict Response
Time Frame: 2.5 months
Population: Due to poor enrollment, data was not analyzed. Adequate data was not collected and the only type of data that remained available was the total # enrolled, some information of the population demographics, and AE/SAE logs that were submitted to the IRB for review.
Arm/Group | Fluoro-L-Thymidine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Fluoro-L-Thymidine: Injection pre-Neoadjuvant Therapy (CRT, CT, or RT) and post-3 weeks Neoadjuvant Therapy (CRT, CT, RT)(3 weeks from the start of Neoadjuvant Therapy) prior to surgery.
  Fluoro-L-Thymidine: 4D-PET/CT imaging with an injection of Fluoro-L-Thymidine at pre-Neoadjuvant Therapy and post-3 weeks Neoadjuvant Therapy prior to surgery.
  Only 5 subjects were followed for AEs/SAEs since one subject withdrew consent prior to any participation in the study.
Arm/Group | Fluoro-L-Thymidine
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoro-L-Thymidine (N=5)
Allergic Reaction to Chemotherapy (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Abnormal Liver Function (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoro-L-Thymidine (N=5)
Abnormal Complete Blood Count (CBC) (Blood and lymphatic system disorders) | 1 (1)
Blood Glucose Level Increased (Endocrine disorders) | 1 (1)
ALT Increased (Hepatobiliary disorders) | 1 (1)
Odynophagia (Ear and labyrinth disorders) | 1 (1)
White Blood Cell (WBC) Count Increased (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment was very slow and poor, resulting in inadequate data collection. As a result, data was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes